CLINICAL TRIAL: NCT00147706
Title: Does Access to an EHR Patient Portal Influence Chronic Disease Outcomes? A Randomised Trial Assessing Clinical and Behavioural Change Outcomes in Patients With CHF, Diabetes, or Secondary CVD
Brief Title: Does Access to an EHR Patient Portal Influence Chronic Disease Outcomes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Nirav Shah, MD, New York University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 051761
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Congestive Heart Failure; Diabetes; Cardiovascular Disease
Keywords: Electronic Health Record; Patient Portal; Chronic Diseases
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Cardiovascular Diseases; Chronic Disease

INTERVENTIONS:
Procedure: Tailored Healthmedia programs on EHR Patient Portal

SUMMARY:
The purpose of this study is to determine if patients with congestive heart failure, diabetes or secondary cardiovascular diseases, who access HealthMedia's online tailored behavior change programs on the electronic health record patient portal have better clinical and behavioral change outcomes.

DETAILED DESCRIPTION:
The specific aims of the study are to determine if e-portal interventions influence:

* Measures of patient activation, patient self-management, treatment adherence, patient satisfaction with care, and disease specific knowledge.
* Process measures relevant to appropriate care for CVD, CHF, and DM.
* Clinical markers of cardiovascular or diabetes morbidity and risk.

These aims will be evaluated in one-year prospective study. Patients who use the portal will be randomized to control (i.e., access to routine portal-related information) and intervention groups (i.e., targeted and periodic messages designed to capture data relevant to self-management; to improve knowledge of their specific disease, tests, and risks; to devise time-dependent goals; and to motivate self-efficacy). Outcomes including activation, satisfaction, and adherence will be measured by telephone interview prior to and one year after intervention, and by lab and clinical measures and data available from the EHR. We will also evaluate potential selection issues among those who sign on to the e-portal by administering the same baseline interview to a matched (by disease and by age) random sample of patients who do not sign on to the e-portal.

Patients with chronic diseases are likely to experience particular benefit from online e-health resources as they have greater information needs and participate in self-management.(Camer, 2000) Unlike traditional office visits, online interactions eliminate the need to travel, are always available and give the patient access to a broad range of information, helping them actively participate in their own care.(Brown, 1999) There is growing evidence that patient education and engagement using e-health applications results in improved patient outcomes in the care of chronic illnesses, improved patient-physician communication, and reduction of anxiety for caregivers.(Brennan et al., 2001; Bronson et al., 1986; Bronson & O'Meara, 1986; Ross et al., 2003a, 2003b) We anticipate demonstrating clinically meaningful improvements in chronic disease health status, using evidence-based science delivered in behaviorally-validated ways.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years or older
* Have medical records in the Geisinger Electronic Health Record
* Have congestive heart failure and/or Diabetes and/or cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
knowledge, behavior change, relevant clinical measures

CONTACTS AND LOCATIONS:
Overall Officials: Walter F Stewart, PhD, Principal Investigator — Geisinger Health Systems; Nirav R Shah, MD. MPH, Study Chair — NYU Langone Health
Locations (1):
- Center for Health Research & Rural Advocacy. Geisinger Clinic, Danville, Pennsylvania, United States